CLINICAL TRIAL: NCT06050135
Title: Roadmap to Parenthood: Testing the Efficacy of a Decision Aid and Planning Tool for Family Building After Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-71534; 1R37CA282148-01 (NIH); NCI-2024-06041 (Registry Identifier: National Cancer Institute Clinical Trials Reporting Program)
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Quality of Life; Parenthood Status
Keywords: Roadmap to Parenthood; Decision aid; Planning tool

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based decision support (Roadmap to Parenthood) (Experimental): Patients will receive access to the Roadmap to Parenthood tool (website). The goal of the Roadmap tool is to encourage young adult females (YA-Fs) to be informed about family-building options, set realistic expectations about potential difficulties, and plan ahead to avoid or mitigate barriers, while also inspiring hope and confidence that parenthood may be achieved, despite their cancer histories.
  Interventions: Other: Roadmap to Parenthood
- Informational booklet (Active Comparator): Patients will receive the web-based Livestrong 'Planning for Life After Cancer: A Guide to Survivorship for Teens and Young Adults' informational booklet, covering many topics (e.g., physical symptoms, emotional concerns, day-to-day needs).
  Interventions: Other: Informational Booklet

INTERVENTIONS:
Other: Roadmap to Parenthood — web-based decision support
  Arms: Web-based decision support (Roadmap to Parenthood)
Other: Informational Booklet — web-based informational booklet about young adult cancer survivorship
  Arms: Informational booklet

SUMMARY:
This study will test a decision support intervention that consists of a web-based 'decision aid and planning tool' for family building after cancer in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth
* Aged 18 to 45 years old
* Understands verbal and written English
* History of a cancer diagnosis.
* Completed cancer treatment(s) with known or uncertain gonadotoxic effects (e.g., systemic chemotherapy, surgery or radiation affecting reproductive organs or hormone regulation, stem cell or bone marrow transplant, and/or immunotherapy)
* Interested in having a future child (or more children) or uncertain about family building plans
* Access to the Internet and use of a computer, tablet, or smartphone
* Ability to understand and the willingness to personally sign the written IRB-approved informed consent document

Exclusion Criteria:

* Currently undergoing cancer treatment excluding long term adjuvant or maintenance therapies, such as tamoxifen
* Significant physical or mental disability that prevents completion of study activities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female cancer survivors
Enrollment: 256 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Decision Conflict Scale | 12 months
  Decisional Conflict Scale is a validated survey that assesses personal uncertainty in making healthcare decisions; modifiable factors contributing to uncertainty; and the quality of the decision made. The survey has 16 questions, with responses on a 5 point scale ranging from "strongly agree" (1) to "strongly disagree" (5). Total scores range from 16 to 80, with higher scores indicating greater uncertainty (worse outcome)

SECONDARY OUTCOMES:
Planning Behaviors for Future Family Building | 12 months
  Yes and No (Y/N) question of whether participants completed "next step" planning behaviors aligned with their family-building goals
Patient-Reported Outcomes Measure-29 (PROMIS-29) Quality of Life | 12 months
  PROMIS-29 assesses seven domains of health-related quality of life including physical function, anxiety, depression, ability to participate in social roles and activities (social participation), fatigue, pain interference, and pain intensity. Items are scored on a 5-point scale (range 1-5). From the sum of the answers to each question in the domain, the total raw score for each domain is calculated, resulting in seven domain scores, each between 4 and 20

OTHER OUTCOMES:
Unmet Fertility Information Needs | 12 months
  The survey has 5 questions, each answered by a Yes / No response. Yes is scored as 1, and no is scored as 0. Total scores range from 0 to 5, with higher scores indicating greater perceived knowledge.
Patient-Reported Outcomes Measure (PROMIS) General Self Efficacy | 12 months
  Questions measures the degree to which people feel confident in managing various situations, problems, and events and confidence in managing negative emotions. Items are scored on a 5-point scale (range 1-5).From the sum of the answers to each question in the domain, the total raw score for each domain is calculated, resulting in seven domain scores, each between 4 and 20
Reproductive Concerns After Cancer (RCAC) Scale | 12 months
  The survey has 18 questions, answered on a 5 point scale ranging from "strongly disagree" (1) to "strongly agree" (5). Total scores range from 18 to 90, with higher scores indicating greater distress (worse outcome).
COMRADE subscale | 12 months
  Items are answered on a 5-point scale from "Strongly Disagree" to "Strongly Agree," with high scores indicating better outcomes
Patient-Reported Outcomes Measure (PROMIS) General Self-Efficacy and Self-Efficacy for Managing Emotions | 12 months
  The PROMIS General Self-Efficacy and Self-Efficacy for Managing Emotions subscales measure the degree to which people feel confident in managing various situations, problems, and events and confidence in managing negative emotions. 21 Questions will assess general self-efficacy in these domains and self-efficacy in managing fertility and family-building issues and emotions. The outcome will be reported as the mean difference from baseline to 1, 6, and 12 months, with standard deviation. Items are answered on a 5-point scale from "Strongly Disagree" to "Strongly Agree," with high scores indicating better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Benedict, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Universtiy, Palo Alto, California, United States